CLINICAL TRIAL: NCT02749812
Title: Beneficial Effects of Obstructive Sleep Apnea Syndrome (OSAS) Treatment by Automatic Continuous Positive Airway Pressure (APAP) vs Constant Continuous Positive Airway Pressure (Constant CPAP) According to the Level of the Efficient Pressure and Its Variability. A Multicentric Randomized Trial
Brief Title: Interest of Treatment of Obstructive Sleep Apnea Syndrome by Constant CPAP and Auto CPAP
Acronym: PREDIVARIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDIVARIUS
Record Dates: First submitted 2016-04-11; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Obstructive Sleep Apnea Syndromes

ARMS (2):
- Constant Continuous Positive Airway Pressure (Experimental)
  Interventions: Device: Constant Continuous Positive Airway Pressure
- automatic Continuous Positive Airway Pressure (Experimental)
  Interventions: Device: Automatic continuous Positive Airway Pressure

INTERVENTIONS:
Device: Constant Continuous Positive Airway Pressure
  Arms: Constant Continuous Positive Airway Pressure
Device: Automatic continuous Positive Airway Pressure
  Arms: automatic Continuous Positive Airway Pressure

SUMMARY:
The investigators propose a multicentric controlled randomized trial whose goal is to evaluate the possibility of a prediction of the efficiency of APAP (automatic continuous positive airway pressure) and constant CPAP (constant positive airway pressure) in 800 severe obstructive sleep apnea syndrome (OSAS) patients according to their profile of pressure variability.

DETAILED DESCRIPTION:
Multicenter open randomized clinical trial involving 800 patients with severe OSAS. After inclusion in the study, the patients will be proposed to initiate CPAP at home (ResMed S9 or PHILIPS PR1) using systematically an APAP mode between wide range of pressure variations (4 to 20 cm H2O) during the first 7day-period of time. After this first period of treatment, an analysis of the report will be released from the APAP in order evaluate the residual AHI, the duration of CPAP use and the amount of leaks in order to confirm CPAP efficiency and observance. Pressure parameters (efficient pressure and variability) will be collected. After randomization according to the further mode of ventilation to use (APAP vs constant CPAP), the patients will be treated at home for 3 months. In the constant CPAP group, efficient pressure will be determined as the P95 (ResMed) or the P90 (PHILIPS) as recommended by the manufacturers, while in the APAP group, the patients will be treated within the same range of pressure variations than during the first 7 day-period. Clinical and polygraphic evaluation will be done after 3 months of treatment, using the combined criteria previously described. In each group, results will be considered according to the efficient pressure value and its variability that were evaluated at the end of the first 7 day-period of treatment

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 with severe OSAS (AHI > 30/h)
* Patients naive of any previous OSAS treatment
* Written informed consent

Exclusion Criteria:

Patients

* with more than 20% of central events at the initial polygraphic recording
* previously treated by CPAP
* previously treated for OSAS by any surgical procedure involving upper airways
* < 18
* with cardiac insufficiency
* with Chronic Obstructive Pulmonary Disease or obesity-hypoventilation syndrome
* without health insurance
* pregnant or lactating
* presumed uncooperativeness or legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
A combined score that takes into account the residual apnea hypopnea index (AHI) under CPAP associated with the value of the Epworth score after 3 months of treatment. | 3 months
  The main objective of this study is to evaluate the ability to predict the mode of CPAP to use (APAP vs constant CPAP) in the treatment of OSAS patients, according to their own level of efficient pressure and its variability obtained on CPAP report after the first 7 days of use in an initial and systematic APAP mode. This prediction will be evaluated by using the association of the residual AHI value under CPAP and the Epworth score value obtained after 3 months of treatment, in each group of CPAP mode (constant vs APAP) used during the study. This combined criteria will be used according an ordinal scale with six levels of severity. It will be evaluated in each group (constant CPAP vs APAP) according to the level of P90 or P95 and the degree of pressure variability obtained during the first 7 day-period of use.